CLINICAL TRIAL: NCT07045480
Title: Prevention of Pressure Ulcers by Effleurage With RIVADOUCE VEGETABLE SKINCARE OIL in Patients at Risk of Pressure Ulcers: Observational Study
Brief Title: Prevention of Pressure Ulcers by Effleurage With RIVADOUCE VEGETABLE SKINCARE OIL in Patients at Risk of Pressure Ulcers
Status: Recruiting | Type: Observational
Sponsor: Laboratoires RIVADIS (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-A01643-44
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Pressure Ulcer Prevention
Keywords: Effleurage; Pressure Ulcer; Topical Emollient; Post-Market Clinical Follow-Up; Rivadouce
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rivadouce Group: Patients aged 18 years and older, at risk of developing pressure ulcers (Braden Scale <18), without existing ulcers at baseline, and for whom RIVADOUCE VEGETABLE SKINCARE OIL is applied via effleurage as part of routine clinical practice. Patients are followed for 35 ± 5 days to monitor the incidence of pressure ulcers and adverse events.

SUMMARY:
This is a prospective, non-interventional, multicenter, post-market clinical follow-up (PMCF) study conducted in real-life conditions to assess the clinical performance and safety of RIVADOUCE VEGETABLE SKINCARE OIL in the prevention of pressure ulcers (PUs) in at-risk adult patients. The product is intended to be applied through effleurage (gentle manual application without pressure) to pressure-prone skin areas as part of standard pressure ulcer prevention protocols.

A total of 252 adult patients, with a Braden Scale score <18 and no existing pressure ulcers at baseline, will be included across 10 to 20 French healthcare centers (e.g., rehabilitation units, long-term care facilities, or nursing homes). Participants will be followed for 35 ± 5 days.

The primary endpoint is the proportion of patients developing at least one stage 1 or higher pressure ulcer (per NPUAP 2014/2019 classification) on treated areas (e.g., sacrum, heels, ischial and trochanteric regions). Secondary endpoints include the time to onset, progression of any developed ulcers, adverse events (AEs), device-related adverse events, and product usage compliance.

This PMCF study is required for the renewal of CE certification under the EU Medical Device Regulation (MDR) 2017/745, and is designed according to ISO 14155:2020 standards. The study will provide updated clinical evidence on the device's safety and performance within its intended use.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of inclusion.
* At risk of developing pressure ulcers, as determined by clinical judgment and a Braden Scale score <18.
* No existing pressure ulcer at the time of inclusion.
* Informed consent signed by the patient, or by a trusted third party or legal representative (for protected adults), after being informed about the study.
* Expected length of stay ≥ 35 days ±5 days in the participating facility.
* Planned use of RIVADOUCE VEGETABLE SKINCARE OIL on one or more pressure-prone areas as part of the facility's standard pressure ulcer prevention protocol.

Exclusion Criteria:

* Use or planned use of multilayer dressings on the pressure-prone areas to be treated with the study product.
* End-of-life patients, defined as having an estimated life expectancy of less than 3 months.
* Patients who are not covered by social health insurance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult patients (≥18 years) who are at risk of developing pressure ulcers, as defined by clinical assessment and a Braden Scale score of less than 18. Eligible participants must have no existing pressure ulcers at baseline and be expected to remain in the participating healthcare facility (e.g., rehabilitation center, nursing home, or long-term care unit) for at least 35 ± 5 days. Patients will receive RIVADOUCE VEGETABLE SKINCARE OIL as part of routine pressure ulcer prevention care, applied by effleurage to pressure-prone skin areas. The study population is representative of frail, often immobilized individuals in geriatric or rehabilitative settings.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Pressure Ulcers on Treated Areas | Day 0 to Day 35 (±5 days)
  Proportion of patients who develop at least one stage ≥1 pressure ulcer (per NPUAP classification 2014/2019) between Day 0 and Day 35 (±5 days) on areas treated with RIVADOUCE VEGETABLE SKINCARE OIL (e.g., sacrum, ischium, trochanter, heels, elbows, spine).

SECONDARY OUTCOMES:
Time to Onset of First Pressure Ulcer on Treated Areas | Day 0 to Day 35 (±5 days)
  Number of days from baseline (Day 0) to first occurrence of a stage ≥1 pressure ulcer on a treated zone.
Occurrence of Adverse Events Related to the Device | Day 0 to Day 35 (±5 days)
  Assessment of whether the oil was applied according to the protocol-defined frequency, zones, and method (effleurage).

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie MEAUME, PhD, Principal Investigator — Hôpital Rotschild
Locations (1):
- Multiples facilities, Multiple Locations, France

IPD SHARING:
Plan to Share IPD: No